CLINICAL TRIAL: NCT02095561
Title: Study of HPV Self Testing Evaluation in the Province of Jujuy, Argentina
Brief Title: Evaluation of Human Papilloma Virus (HPV) Self-testing to Increase Screening Uptake
Acronym: EMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional del Cáncer, Argentina (Other Government)
Collaborators: Ministerio de Salud de Jujuy (Other Government); International Agency for Research on Cancer (Other); National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Silvina Arrossi, PhD in Demography, National Council of Scientific and Technical Research, Argentina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 01-1CU
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: HPV self testing; screening uptake; cervical cáncer; cervical intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HPV Self testing (Experimental): HPV self testing offered by CHWs during home visits
  Interventions: Other: HPV self testing
- HPV at health centers (No Intervention): Community Health Workers instructed women about cervical cancer and HPV testing and advised them on how to seek screening at health centers.

INTERVENTIONS:
Other: HPV self testing — Community Health Workers instructed women about cervical cancer and HPV testing, advised them on how to seek screening at health centers, and offered them the option of self-testing, providing women with educational materials on how to perform it.
  Arms: HPV Self testing

SUMMARY:
Cervical cancer is a leading cause of mortality among women in developing countries. A key factor has been the failure to achieve good coverage. The development in the last years of HPV-DNA based tests has changed the scenario, because it combines a high performance to detect disease with a reduction of screening frequency. Through self-testing, HPV testing has the potential of reducing social and health service barriers faced by women to access screening.

This study is carried out in Jujuy, one of the Argentinian provinces with highest cervical cancer mortality rates and where HPV testing has been introduced as a primary screening test for all women attending public health sector. The study was conducted between July 2012-December 2013, and supported by the Argentinean National Cancer Institute. The protocol was approved by the institutional review committees of the Ministry of Health of Jujuy.

This trial is a randomized by population clusters study that aims to assess the effectiveness of self-testing to increase coverage. The aims of this study are: a) to assess the self-test effectiveness to increase the participation of women in screening programs, b) to assess the self-test acceptability by women, c) to assess HPV self-test effectiveness measurement for the detection of CIN2+ lesions against cytology in primary screening.

An overall number of 200 community health workers (CHWs) from the Primary Health Care System (PHCS) of Jujuy will be randomized into two groups that will be named Self-test Group (ST) and Conventional Sample Group (CS):

1. ST Group: CHWs will invite eligible women of their area to choose between doing a self-test or having a conventional sample taken by a health professional of the closest health care center.
2. CS Group: CHWs will invite eligible women in their area to have a conventional sample taken by a health care professional of the nearest health care center.

In order to measure the self-test relative sensitivity against cytology to detect CIN2+ in primary screening, all the women in the Self-test Group who have decided to do the self-test and all the women of 30 years of age and older that were screened with cytology by the provincial program for the prevention of cervical cancer in 2011 will be considered.

A database built specifically for the study will be used; it will hold the list of eligible women to participate in the study. The records of women of 30 years of age and older residing in the areas included in the study will be imported from the PHCS databases.

In addition, the data surveyed by the study will be uploaded: randomization Group, presence of the woman at home during the CHW's visit, agreement to participate in the study, realization of self-test (in the corresponding group), and if appropriate, reasons for not doing the self-test. Lastly, the HPV Test realization will be uploaded importing the data on SITAM, (link of data done as from the identity card number).

Data Analysis

Self-test acceptability: Acceptability is defined as the number of women accepting the self-test against the number of women offered the option between the self-test and the conventional sample (proportion of women accepting the self-test). The acceptability in this population will be estimated as the average of acceptabilities calculated by CHW, as to control the impact of the CHWs on acceptability and reach an appropriate variance estimate. Besides, the variability introduced by the CHWs on acceptability will be studied and the results obtained by male and female CHWs will be compared, as well as those obtained by the CHWs in rural and urban areas.

Self-test effectiveness to enhance participation of women in screening and diagnosis: There will be a comparison of the percentage of women that did the HPV test in the Self-test group and the Conventional sample group. Three different coverage indicators will be considered for every CHW. These will be defined as the number of women screened within the field work regarding:

1. The number of women reached by the CHW who accepted participating in the study.
2. The number of eligible women for that CHW (regardless of whether the CHW was able to contact them or not).

The effect of the strategy (offering the self-test option against promotion of the conventional sample) will be estimated for each one of the coverage measures using a means difference test or a non-parametric test for independent samples.

CIN 2+ detection rate: The effectiveness of the HPV Self-test against screening cytology to detect CIN2+ will be estimated as the detection rates difference and as the detection rates ratio. In addition, there will be a comparison of the CIN2+ detection rate in the group of women who did the self-test against the total number of women in the province of Jujuy that were tested for HPV (conventional sample strategy + triage Pap test) until December 2012.

DETAILED DESCRIPTION:
Description of the problem and study rationale

High screening coverage of women at higher risk is an essential component within organized cervical cancer (CC) prevention programs. Yet, reaching high levels of coverage is a challenge, mainly for programs implemented in developing countries that, in most cases, have not achieved high coverage levels to effectively have an impact on the incidence and mortality of the disease1,2.

In Argentina, it is estimated that 40% of poor women have never participated in screening programs3. It has been shown that it is among those women with low screening frequency that cervical cancer is mainly diagnosed4. In our country, the coverage map shows an inverse correspondence with the cervical cancer mortality map. Women living in the Northwest and Northeast regions, where mortality rates are highest, are the most likely to be screening underusers.

The lack of information about CC prevention, the lack of support networks, shame related to sexuality and the body, and fear of cancer are factors that hinder an informed decision-making process by women about their own health care. In turn, the autonomy of women is often conditioned by the characteristics of the health systems responding to a top-down and medicalized system where there is an asymmetry of knowledge and power between health care professionals and users.

Since the discovery of the causal association between oncogenic HPV (Human Papilloma Virus) and CC, new screening HPV detection-based tools have been developed. The hybrid capture HPV test (HC2) detects the presence of DNA of the 13 high oncogenic risk types in the woman's cervix. It's been proved that the HPV test is highly effective for the detection of pre-cancerous lesions and reduction of cervical cancer mortality5.

In the province of Jujuy CC HC2 is available in all public health centers since 2011, with the aim of improving the effectiveness in the detection of high-grade lesions and cancer and reduce mortality rates.

One of the challenges for programs introducing HPV testing is to continue improving the screening coverage indicators. This new technology has the potential to reduce screening access barriers, given the fact that the HPV test allows for self-testing, a practice that can be done at home. With the self-test the woman collects herself a vaginal sample with a brush used for that purpose.

Studies carried out in different countries of the world and Latin America have shown that the HPV self-test acceptability is high6. The vaginal self-test allows to overcome some of the barriers associated with screening such as geographical accessibility and shame of having a sample taken by a health professional. That is, the self-test has a big potential to increase screening coverage, allowing women enhanced autonomy for their cervical cancer prevention care.

The HC2 HPV test is a molecular biology technology that detects the presence of 13 high oncogenic risk DNA types (16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, and 68) in the cervix cells. It is an accurate technology, highly reproducible and with an estimated sensitivity of more than 90%, much higher than the cytology. Different studies in Latin America and the world account for the HPV Test higher sensitivity against cytology7,8,9,10,11,12,13,14.

At the same time, the HC2 HPV test is the only one in the world whose effectiveness to reduce cervical cancer incidence and mortality has been scientifically proved. A study conducted in India15 concluded that the rates of incidence and mortality were significantly higher within the groups screened with cytology or visual inspection with acetic acid (VIA) as compared to the group screened with HC2. HC2 test screening was able to reach a reduction of almost 50% in the mortality rate.

As far as the self-test, its higher sensitivity against cytology for the detection of cervix cancer precursor lesions (CIN2+) was also observed in various studies11,16.

The CIN2+ detection rate (histologically confirmed diagnosis) also shows a relative advantage of the HPV test over cytology. Different studies have found that detection of CIN2+ is higher in the case of the self-test against cytology 17,18. On the other hand, a study carried out in Mexico found that the CIN2+ lesions self-test detection rate is 3.4 times higher over that of cytology (relative sensitivity)19.

Setting of the study

The province of Jujuy was selected to develop this study due to the fact that screening based on HPV testing as a primary test was introduced in 2011. The province of Jujuy has a high mortality rate (11.8 x 100.000 women over the 2008-2011 period) and it is one of the provinces set as a priority in the National Program for the Prevention of Cervical Cancer. The Primary Health Care System (PHC) integrates approximately 700 CHWs that once a semester visit approximately 110.000 households. In each visit, CHWs contact adults in the household and perform health-related tasks including promotion of cervical cancer screening. CHW's performance is evaluated annually and classified as good or regular.

Goals of the study

A cluster randomized trial will be conducted; it will include a total number of 150-200 community Health Workers (CHWs) and 6.000 women.

The aim of this study is:

1. to assess the self-test effectiveness to increase the participation of women in screening programs,
2. to assess the self-test acceptability by women.
3. to assess HPV self-test effectiveness for detection of CIN2+ lesions against cytology in primary screening.

Study randomized by population clusters

An overall number of 150-200 CHWs from the Primary Health Care System (PHCS) of the Province of Jujuy will be randomized into two groups: Self-test Group (ST) and Conventional Sample Group (CS)

1. ST Group: CHWs will invite eligible women of their area to choose between doing a self-test or having a conventional sample taken by a health professional at the closest health care center.
2. CS Group: CHWs will invite eligible women in their area to have a conventional sample taken by a health care professional at the nearest health care center.

1) Procedures to carry out in each group:

1.1) Active search

• Self-test Group:

During the home visits that CHWs carry during health rounds, selected CHWs will visit every household they are in charge of and will invite eligible women to participate in the study, providing them with the necessary information about the goals and activities involved. Eligible women willing to participate in the study will be invited to sign an informed consent. Next, they will be offered the possibility of doing a self-test or to visit a health care center to have a sample taken by a health care professional. Women who agree on the self-test will be given the option to have more time to do the test if they need so and the CHWs will come back later to pick up the collecting tube. CHWs will explain the procedure based on the communication material designed for that purpose. Women who decide to be screened at health care centers will receive information about available timetables. The CHWs will bring the self-taken sample to the health care center, where all collecting tubes will be stocked to be sent to the provincial HPV laboratory, according to usual procedures and delivery schedules.

CHWs will update the F883 template, the standard PHC form used by CHWs to collect socio-demographic and health data of the household and its members. In addition to that, CHWs will use a specific questionnaire to collect basic about inclusion/exclusion criteria, self-testing acceptability and reasons for doing/not doing self-testing.

• Conventional Sample group:

During the home visits that CHWs carry during health rounds, selected CHWs will visit every household they are in charge of and will invite the eligible women to participate in the study, providing them with the necessary information about the goals and activities involved. Eligible women willing to participate in the study will be invited to sign an informed consent. Next, they will be given an education talk promoting cervical screening. They will be given information about HPV testing at health care centers as well as educational material on the prevention of the disease.

CHWs will update the F883 template, the standard PHC form used by CHWs to collect socio-demographic and health data of the household and its members. In addition to that, CHWs will use a specific questionnaire to collect basic about inclusion/exclusion criteria,

Women from this group, upon visiting the health care center for the conventional test, will be taken an HPV and Pap test at the same time, based on the provincial protocols and regulation framework. Samples will be sent to be read at the Cytology and HPV Laboratory, according to standard provincial mechanisms.

1.2) Delivery of results, follow up and treatment:

• Self-test group:

Women tested HPV positive will receive the visit of the CHW to inform them of the result. They will be invited to undergo diagnosis studies (colposcopy/biopsy) at their closest health care center. The CHW will brief them on the availability of timetables, professionals and health care centers.

Those women with suspicious colposcopic images will have a targeted colposcopy-directed biopsy taken, to be read by the provincial pathological anatomy laboratory.

Women with histologically confirmed precancerous lesions wil be followed up and treated based on the protocols established on the Recommendations for screening, follow up and treatment of women for the prevention of cervical cancer in the framework of the HPV test incorporation, by the National Ministry of Health20.

The data about Pap tests, colposcopy, biopsy and treatments will be registered at SITAM (screening information system), following the Provincial Program for Cervical Cancer Prevention regulation.

• Conventional sample group:

Women tested HPV positive, with abnormal Pap test, will be visited by the CHW to inform them of the result and invite them to undergo a colposcopy at their closest health care center. The CHW will brief them on the availability of timetables, professionals and health care centers.

Women tested HPV positive but with a normal Pap test, will receive the results based on the usual procedures set forth by the Provincial Program for the Prevention of Cervical Cancer.

Those women with suspicious colposcopic images will have a targeted colposcopy-directed biopsy taken, to be read by the provincial pathological anatomy laboratory.

Women with a histologically confirmed precancerous lesion should be followed up and treated based on the protocols set forth in the Recommendations for screening, follow up and prevention of cervical cancer in the framework of the HPV test incorporation, by the National Ministry of Health20.

The data about Pap tests, colposcopy, biopsy and treatments will be registered in SITAM, based on the Provincial Program for the Prevention of Cervical Cancer regulation.

2. Training for CHWs:

All participating CHWs will be informed about the study and a special training will be provided. During the training sessions, the goals of the study, the main activities to be carried out and the specific tasks that each one of them will have to perform will be explained.

3. Production of communications material:

Informative material will be prepared for CHWs participating in the study, the main goals of the study will be explained in it and guidelines with the steps to follow during the home visit will be provided to them.

Similarly, a special leaflet will be prepared with the self-test instructions to be delivered to those women to whom that option is offered.

Besides, all contacted women will be given general leaflets on cervical cancer prevention and the HPV Test and those women that did the self-test will be given a leaflet on the meaning of HPV Test results.

4. Sample selection and size

1. Proposed sample size for the coverage study

   With the purpose of selecting CHWs participating in the study, a list of all the CHWs of the province of Jujuy will be made (N = 678). Then they will be classified by gender and type of health care center (urban or rural). The CHWs that over the year 2011 have been rated of regular performance by the PHC system will be excluded from the study.

   150-200 CHWs will be randomly selected, in a sample proportional to the size of four strata defined by gender and health care center type. The CHWs selected in every stratum will be randomly allocated to each one of the study groups (half for the Self-test group and half for the Conventional Sample group).

   Assuming that a CHW will enroll an average of 40 women (with a minimum target of 20 women) in the two visits of the round, the overall number of women enrolled in every study group will approximately be at least 75 x 40 = 3.000 (number of CHWs x number of women per CHW) with a total number of 6.000 women in the study. We assume that the coefficient of intra-class correlation (CIC) is 0.05, 0.075 or 0.10 the power to detect a 10% change (from 50% to 60%) in the first coverage indicator for a 5% level of significance test is 0.999, 0.97 and 0.93 respectively.
2. Self-test acceptability estimate

   Acceptability is defined as the percentage of women accepting doing the self-test against the number of women offered the self-test or the conventional sample option. Under the scenario described in the previous section the expected half-length of the 95% confidence interval for acceptability within the population is 3.1%, 3.5% and 4.0% for a CIC of 0.05, 0.075 and 0.1 respectively.

   These values are dawned considering the worst situation regarding the length of the confidence interval, which stems from assuming an acceptability of 50%.
3. Sample size for the CIN2+ detection rate comparison of the HPV Self-test versus cytology as a primary screening method

We will compare the detection rate of histologically confirmed CIN2+ lesions diagnosed in 2011 within the framework of the provincial program for the prevention of cervical cancer, based on cytology as primary screening method, against the HPV Self-test detection rate (relative sensitivity). This analysis will include approximately 20.000 women of 30 years of age and older screened with cytology during the year 2011, in the framework of the provincial screening program, and the 3.000 women that are expected to be screened by means of the HPV Self-test within the framework of the present research project.

The cytology detection rate for the year 2011 in the province of Jujuy is of approximately 0.8%. If it is assumed that with the HPV Self-test the detection rate to be reached will be of 1.4%, 1.6%, 1.8% or 2.0%, the power of the one-tailed test (5% level of significance) to compare the CIN2+ detection rates turns out to be 0.895, 0.977, 0.966 and 0.999 respectively. The power calculation was done assuming there is no impact produced by the CHW on the CIN2+ detection rate.

5. Database:

A database built specifically for the study will be used; it will include data about randomization Group, agreement to participate in the study, basic socio-demographic data, realization of self-test (in the corresponding group), and if appropriate, reasons for doing/not doing the self-test. Finally, the HPV Test realization will be uploaded importing the data from SITAM, linking data based on the Unique Identification Number (DNI).

Data entry will be done through specific software that will include range and inter-item consistency checks. Entries out of the expected range will not be allowed. Data entry will be done by 3 data enters, with re-entry of 20% of questionnaires for quality control. Data will be stored in files (TXT, DBF, SQL) compatible with their analysis with statistical packages (Stata).

The data cleaning process will actively search for errors in a planned way. Data screening will include searching for four types of oddities: outliers (including inconsistencies), strange patterns in distributions, and unexpected analysis results. Screening methods will include browsing of data tables after sorting, printouts of variables not passing consistency checks, graphical exploration of distribution, frequency distributions and cross-tabulations and summary statistics. Once errors have been identified, we will go to previous stages of the data flow to see whether the value is consistently the same. If no error is found in the data entry phase, we will question the interviewer about what may have happened. If possible, we will contact the interviewee for repeated measurement.

Accuracy of previous HPV test reported by the woman will be crossed with information from the laboratory database (SITAM). Those women having reported not having a previous HPV test, but with a test in the SITAM data base will be excluded from the study.

The project database will be also matched with the PHC database. For that purpose, the records of women of 30 years of age and older residing in the areas included in the study will be imported from the PHCS databases, including name, DNI and basic socio-demographic data of the woman.

Plan for missing data

Data are exhaustive and complete for all samples arriving to the HPV laboratory. Because we define the outcomes as number of tests effectively recorded in the laboratory database (SITAM)/ number of women in the study arm, we do not expect to have missing data in the main outcome.

SITAM database is less complete regarding follow-up diagnosis procedures: colposcopy and biopsies. In those cases where HPV+ women have missing data for colposcopy and/or biopsy results, the project team will contact Navigators from the Provincial Program for Cervical Cancer Prevention. Usual navigators´ role in the provincial Program is to contact women with abnormal results that have had problems to complete diagnosis/treatment procedures to provide them support so they can be able to finish the process. They can also contact health professionals to verify information reported by women: for example, in cases where women reported having been treated but no data is registered in SITAM. In that case, they contact the health professional to verify treatment provided and its results. Information gathered by navigators is entered in SITAM in a specific module which will be also used to complete data for missing cases.

6. Data analysis:

Data analysis will be done through specific commercial softwares (STATA 10.0 or SAS).

6.1 Self-test acceptability:

Acceptability is defined as the number of women accepting the self-test against the number of women offered the option between the self-test and the conventional sample (proportion of women accepting the self-test). Although all CHWs will receive the same instructions and material, it is to be expected that there will be differences in the way the self-test is offered, be it because they are more convinced about the relative advantages, or for their gender condition, etc. The acceptability in this population will be estimated as the average of acceptabilities calculated by CHW, as to control the impact of the CHWs on acceptability and reach an appropriate variance estimate. Besides, the variability introduced by the CHWs on acceptability will be studied and the results obtained by male and female CHWs will be compared, as well as those obtained by the CHWs in rural and urban areas.

6.2 Self-test effectiveness to enhance participation of women in screening and diagnosis:

There will be a comparison of the percentage of women that did the HPV test in the Self-test group and the Conventional sample group. Three different coverage indicators will be considered for every CHW. These will be defined as the number of women screened within the field work regarding:

1. The number of women reached by the CHW who accepted participating in the study.
2. The number of eligible women for that CHW (regardless of whether the CHW was able to contact them or not).

For every CHW we will measure the adherence to the indication of follow up diagnosis as well as the number of women with colposcopy indication that underwent a colposcopy within the follow-up period over the overall number of women with colposcopy indication.

The effect of the strategy (offering the self-test option against promotion of the conventional sample) will be estimated for each one of the coverage measures using a means difference test or a non-parametric test for independent samples.

6.3 CIN 2+ detection rate:

The effectiveness of the HPV Self-test against screening cytology to detect CIN2+ will be estimated as the detection rates difference and as the detection rates ratio. Specific estimates will be provided as well as intervals of confidence for both measures of effectiveness and accurate or asymptotic tests will be performed as appropriate based on the number of CIN2+ detected.

In addition, there will be a comparison of the CIN2+ detection rate in the group of women who did the self-test against the total number of women in the province of Jujuy that were tested for HPV (conventional sample strategy + triage Pap test) until December 2012. The power of the comparison for the difference observed will be informed upon reporting the results.

ELIGIBILITY:
Inclusion Criteria:

* woman aged 30 or older
* lived in a household visited by one of study CHWs

Exclusion Criteria:

* hysterectomy
* been treated for a precancerous lesion
* with previous HPV test
* pregnant
* mentally-disabled.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6013 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvina Arrossi, PhD, Principal Investigator — National Council of Scientific and Technical Research, Argentina
Locations (1):
- Instituto Nacional Del Cáncer, Argentina, Ciudad de Buenos Aires, Argentina

REFERENCES:
- [Derived] Arrossi S, Thouyaret L, Herrero R, Campanera A, Magdaleno A, Cuberli M, Barletta P, Laudi R, Orellana L; EMA Study team. Effect of self-collection of HPV DNA offered by community health workers at home visits on uptake of screening for cervical cancer (the EMA study): a population-based cluster-randomised trial. Lancet Glob Health. 2015 Feb;3(2):e85-94. doi: 10.1016/S2214-109X(14)70354-7. PMID 25617202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPV Self Testing | HPV at Health Centers
Started | 3049 | 2964
Self-testing Acceptability | 2616 | 0 (Acceptablity only applies to the group of women being offered self-testing.)
HPV Self-tested Women | 2519 | 0 (HPV self-testing only applies to the HPV self-testing arm)
HPV Tested at Health Centers | 99 | 599
Completed | 3049 (All women are part of the study, independently of whether they were tested or not.) | 2964 (All women are part of the study, independently of whether they were tested or not.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HPV Self Testing | HPV at Health Centers | Total
Number analyzed (Participants) | 3049 | 2964 | 6013
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2840 | 2787 | 5627
  >=65 years | 209 | 177 | 386
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3049 | 2964 | 6013
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 3049 | 2964 | 6013
Education Level [Number; unit: participants]
  Never went to school/Primary (incomplete) | 488 | 472 | 960
  Primary (complete)/Secondary (incomplete) | 1373 | 1291 | 2664
  Secondary complete | 600 | 593 | 1193
  Tertiary (incomplete/complete) | 401 | 381 | 782
  Missing cases | 187 | 227 | 414
Health insurance [Number; unit: participants]
  Public system | 1472 | 1555 | 3027
  private/social security | 1409 | 1241 | 2650
  Missing cases | 168 | 168 | 336
Pap test in last four years [Number; unit: participants]
  Yes | 889 | 838 | 1727
  No | 2160 | 2126 | 4286

OUTCOME MEASURES:

1. Primary Outcome: Screening Uptake
Description: The primary outcome was screening uptake, defined as: a) the proportion of participant women with any HPV test (self-test or HPV at health centers) in the information system, in the 6 months after the CHW visit, and b) the proportion of women in the intervention group with a self-test in SITAM, in the same 6 month period.
Time Frame: within 6 months after the intervention
Measure: Number; unit: participants
Arm/Group | HPV Self Testing | HPV at Health Centers
Number analyzed (Participants) | 3049 | 2964
participants
  Self-tested women | 2519 | 0
  HPV-tested | 2618 | 599

2. Secondary Outcome: Acceptability
Description: Defined as the proportion of women from the intervention group who were offered self-testing and accepted, as documented in the questionnaire, independently of if they ended up with a test in the information system.
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | HPV Self Testing | HPV at Health Centers
Number analyzed (Participants) | 3049 | 2964
participants | 2616 | 0

3. Secondary Outcome: CIN2+ Detection Rate
Description: calculated as the percentage of women with histologically confirmed CIN2+ over total number of tested women, both for women with self-testing and those HPV tests taken at health centers.
Time Frame: within one year after the CHW visits
Population: Population included in the HPV self-testing group to calculate CIN2+ detection rate includes only women who were self-tested (n=2519). It excludes 99 women from this group who were not self-tested and were tested at health centers.
Measure: Number; unit: percentage of CIN2+/ women screened
Arm/Group | HPV Self Testing | HPV at Health Centers
Number analyzed (Participants) | 2519 | 599
percentage of CIN2+/ women screened | 1.15 | 1.17

4. Secondary Outcome: HPV Positivity
Description: Calculated as the percentage of women with positive HPV test over total number of tested women, both for women with self-testing and those HPV tests taken at health centers.
Time Frame: within 6 months after the CHW visits
Population: Population included in the HPV self-testing group to calculate positivity includes only women who were self-tested (n=2519). It excludes 99 women from this group who were not self-tested and were tested at health centers.
Measure: Number; unit: percentage of positive tests/tested wome
Arm/Group | HPV Self Testing | HPV at Health Centers
Number analyzed (Participants) | 2519 | 599
percentage of positive tests/tested wome | 11.8 | 11.9

ADVERSE EVENTS:
Time Frame: Overall study period
Arm/Group | HPV Self Testing | HPV at Health Centers
Serious Adverse Events (participants affected / at risk) | 0/3049 | 0/2964
Other Adverse Events (participants affected / at risk) | 0/3049 | 0/2964

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No